CLINICAL TRIAL: NCT01358123
Title: Von Willebrand Factor As Non-Invasive Predictor Of Clinically Significant Portal Hypertension And Mortality In Patients With Liver Cirrhosis
Brief Title: Value of Von Willebrand Factor in Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arnulf Ferlitsch, MD, Associate Professor, Medical University of Vienna
Other Study IDs: vwfcirr
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: liver cirrhosis; portal hypertension; survival; von willebrand factor; hepatic venous pressure gradient
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In patients with liver cirrhosis elevated levels of von Willebrand factor antigen (vWF-Ag) are found frequently but the clinical significance is unclear. vWF-Ag plays an important role in primary haemostasis and development of thrombotic vascular obliteration is discussed as a possible mechanism leading to portal hypertension. Invasive measurement of hepatic venous pressure gradient (HVPG) is the current gold standard for the diagnosis of portal hypertension. The investigators hypothesize that vWF-Ag levels in plasma may correlate with portal pressure and predict clinically significant portal hypertension (CSPH, HVPG >=10mmHg) and its complications.

DETAILED DESCRIPTION:
Patients with alcoholic, viral (chronic hepatitis C), and cryptogenic liver cirrhosis are included. Portal hemodynamics are assessed by HVPG measurement, vWF-Ag levels were measured by ELISA. Results will be compared. 3 and 6 months mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis

Exclusion Criteria:

* no HVPG measurement

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis of all etioloiges, routinely scheduled for routine HVPG measurement will systematically be included during the study period
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
von Willebrand Factor Ag Level | at first visit (HVPG Measurement) (day 1)
  von Willebrand Factor Antigen Levels are measured via ELISA and compared /corrlated to Hepatic Venous Pressure Gradient (HVPG). von Willebrand Factor Antigen levels are drawn and analyzed at the day of HVPG measurement. No follow up measurements will be performed, survival will be measured as secondary outcome parameter

SECONDARY OUTCOMES:
Overall Mortality | 3 Months
  Survival of Patients after index measurement of von Willebrand Factor and HVPG

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria